CLINICAL TRIAL: NCT03732430
Title: A Safety and Efficacy Study of CT-Guided Adaptive Radiation Therapy With Anti-PD-1 Antibody Adjuvant Immunotherapy in Patients With Thoracic Cancer (CARTAI)
Brief Title: CT-Guided Adaptive Radiation Therapy Combine With Anti-PD-1 Antibody Adjuvant Immunotherapy for Thoracic Cancer Patients
Acronym: CARTAI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, Head of Department of Radiation Oncology, Chief Physician, Taizhou Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YHH-201811
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Thoracic Malignancies
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-PD-1 antibody (Experimental): IBI308 200mg intravenous drip every three weeks following adaptive radiation therapy.
  Interventions: Drug: IBI308

INTERVENTIONS:
Drug: IBI308 — A humanized anti-PD-1 monoclonal antibody

SUMMARY:
This phase II study is to evaluate the safety and efficacy of CT-based adaptive radiation therapy followed by adjuvant anti-PD-1 antibody immunotherapy in treating patients with different types and stages of thoracic malignancies. (CARTAI)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity of anti-programmed cell death 1 (PD-1) inhibition consolidation therapy after radiation therapy for multiple thoracic malignancies.

SECONDARY OBJECTIVES:

I. To assess the efficacy of adjuvant anti-PD-1 antibody immunotherapy after radiotherapy.

II. To understand the dynamics and interactions of IDO with others immune pathway biomarkers.

III. To evaluate whether IDO immune status could predict the treatment outcomes of radiation and immune combined therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed inform consent form
2. Age >= 18 years and <= 75 years
3. Histologically or cytologically confirmed advanced/metastatic thoracic malignancies
4. Patients must receive adaptive radiation therapy within 45 days before the first dose of trial treatment
5. Eastern Cooperative Oncology Group performance status of 0 or 1
6. Life expectancy >= 8 weeks
7. Adequate hematologic and end organ function

Exclusion Criteria:

1. Prior exposure to any immune checkpoint inhibitors including but not limited to anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibodies.
2. Prior exposure to any other thoracic radiation therapy before this time radiation therapy.
3. Prior exposure to steroid therapy or any other form of immunosuppressive therapy within 14 days before the first dose of trial treatment
4. No active second cancers
5. Active or prior autoimmune disease or immunodeficiency.
6. Active infections including but not limited to hepatitis B, C ,and HIV.
7. Significant cardiovascular disease
8. Active or untreated central nervous system (CNS) metastases
9. Any unresolved toxicity CTCAE >= Grade 3 from the prior radiation therapy.
10. Known hypersensitivity to humanized antibodies or fusion proteins or any of study drug excipients.
11. Known psychiatric or physical impairments that would interfere with cooperation with the protocol of this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
AEs and SAEs at 6 months | 6 months
  Number of participants with adverse events and serious adverse events at 6 months will be measured. [CTCAE v4.03]

SECONDARY OUTCOMES:
ORR | Estimated to be up to 3 years
  Objective response rate is the percentage of patients with at least once occurrence of PR or CR [RECIST v1.1]
DoR | Estimated to be up to 3 years
  Duration of response is the time interval from first occurrence of PR or CR until PD or death [RECIST v1.1]
AEs | Estimated to be up to 3 years
  Number of patients with acute and chronic adverse events will be measured [CTCAE v4.03]
PFS | Estimated to be up to 3 years
  Progression-Free-Survival is the time interval from the start of treatment until disease progression or death by any cause [RECIST v1.1]
OS | Estimated to be up to 3 years
  Overall Survival is the time interval from the start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Fengming (Spring) Kong, MD, Principal Investigator — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University; Haihua Yang, MD, Principal Investigator — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University; Yinnan Meng, MD, Principal Investigator — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Locations (1):
- Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No